CLINICAL TRIAL: NCT01508988
Title: A Double-masked Placebo-controlled, Single Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ONO-9054 in Healthy Adult Subjects
Brief Title: Single Dose Escalation Study of ONO-9054 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharma USA Inc (Industry)
Responsible Party: Sponsor
Organization: Ono Pharmaceutical Co. Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-9054IOU001
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Healthy Adult Subjects
Keywords: ONO-9054; adult healthy volunteers; single dose; phase 1
MeSH Terms: interventions — propan-2-yl 4-(6-(4-(2,5-difluorophenoxy)-3-hydroxybut-1-en-1-yl)-7-hydroxyoctahydro-2H-cyclopenta(b)oxepin-3-yl)butanoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Eye drops 0.3 µg/mL (Experimental)
  Interventions: Drug: ONO-9054
- Eye drops 1 µg/mL (Experimental)
  Interventions: Drug: ONO-9054
- Eye drops 3 µg/mL (Experimental)
  Interventions: Drug: ONO-9054
- Eye drops 10 µg/mL (Experimental)
  Interventions: Drug: ONO-9054
- Eye drops 20 µg/mL (Experimental)
  Interventions: Drug: ONO-9054
- Eye drops 30 µg/mL (Experimental)
  Interventions: Drug: ONO-9054
- Eye drops placebo (Experimental)
  Interventions: Drug: ONO-9054

INTERVENTIONS:
Drug: ONO-9054 — Eye drops 0.3 µg/mL both eyes on Day one
  Arms: Eye drops 0.3 µg/mL
Drug: ONO-9054 — Eye drops 1 µg/mL both eyes on Day one
  Arms: Eye drops 1 µg/mL
Drug: ONO-9054 — Eye drops 3 µg/mL both eyes on Day one
  Arms: Eye drops 3 µg/mL
Drug: ONO-9054 — Eye drops 10 µg/mL both eyes on Day one
  Arms: Eye drops 10 µg/mL
Drug: ONO-9054 — Eye drops 20 µg/mL both eyes on Day one
  Arms: Eye drops 20 µg/mL
Drug: ONO-9054 — Eye drops 30 µg/mL both eyes on Day one
  Arms: Eye drops 30 µg/mL
Drug: ONO-9054 — Matched-placebo eye drops dosed in the same manner as ONO-9054 in both eyes on Day one
  Arms: Eye drops placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of ascending single doses of ONO-9054 administered as a single drop in healthy adult subjects. The secondary objectives are to characterize the pharmacokinetic (PK) profile of ONO-9054 and its metabolite in plasma and to evaluate the pharmacodynamic (PD) profile.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects, aged 18-64 inclusive
* Body mass index (BMI) of 19-35 kg/m2 (inclusive)
* IOP measurement oculus uterque (OU, both eyes) < 21 mm Hg (inclusive) at screening and Day -1
* Best corrected visual acuity (BCVA) 20/30 or better (Snellen Equivalent) at both the screening visit and Day -1

Exclusion Criteria:

* Any history of severe ocular trauma in either eye at any time
* Any history of previous intraocular or ocular laser surgery within the past 3 months or any refractive surgery procedure within the past 6 months of the screening visit in either eye
* Current or chronic history of ocular infection within the past 3 months of screening visit in either eye OR ongoing or recurrent ocular inflammation in either eye
* At the ophthalmic investigator's discretion, any subjects who have a history of any significant ocular conditions in either eye that would contraindicate the use of the study medication, or that might affect the study conduct, or the interpretation of the study results
* Use of any non-diagnostic topical ophthalmic solutions except for sponsor-recommended tear substitutes from admission to the study unit through the duration of the study
* History of clinically significant drug or food allergy, positive HIV, hepatitis B or C at screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ONO-9054 using vital signs, ECGs, laboratory tests, ocular exams, spirometry, physical examinations and incidence/severity of adverse events | up to 4 days

SECONDARY OUTCOMES:
1. Characterization of PK profiles of ONO-9054 and metabolite through measurement of drug concentration in plasma sample | up to 2 days
2. Pharmacodynamic evaluation of ophthalmic effects by measuring the degree and duration of intraocular pressure lowering | up to 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Ono Pharma USA, Inc., Study Director — Ono Pharmaceutical Co. Ltd
Locations (1):
- Covance Phase 1 Unit, Dallas, Texas, United States

REFERENCES:
- [Derived] Suto F, Rowe-Rendleman CL, Ouchi T, Jamil A, Wood A, Ward CL. A Novel Dual Agonist of EP3 and FP Receptors for OAG and OHT: Safety, Pharmacokinetics, and Pharmacodynamics of ONO-9054 in Healthy Volunteers. Invest Ophthalmol Vis Sci. 2015 Dec;56(13):7963-70. doi: 10.1167/iovs.15-18166. PMID 26720443